CLINICAL TRIAL: NCT02460081
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled, Dose Range Finding Study to Evaluate the Safety, Hemodynamic Effects and Efficacy of Intramuscular Injection of Human Placenta-derived Cells (Pda-002) in Subjects Who Have Diabetic Foot Ulcer With Peripheral Arterial Disease
Brief Title: Safety, Hemodynamic Effects and Efficacy of Intramuscular PDA-002 in Subjects Who Have Diabetic Foot Ulcer With Peripheral Arterial Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinued due to significant delays in the expected availability of data.
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-PDA-002-DFU-003
Record Dates: First submitted 2015-04-21; First posted 2015-06-02 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2016-04

CONDITIONS: Diabetic Foot; Peripheral Arterial Disease
Keywords: PDA-002; Diabetic Foot Ulcer; Peripheral arterial disease; Phase 2; Randomized
MeSH Terms: conditions — Diabetic Foot; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PDA-002 -3x10^6 cells (Experimental): Subjects will be treated with Investigational Product (IP) administered intramuscular (IM) on Study Days 1, 29 and 57.
  Interventions: Drug: PDA-002
- PDA-002 - 30X10^6 cells (Experimental): Subjects will be treated with IP administered IM on Study Days 1, 29 and 57.
  Interventions: Drug: PDA-002
- Placebo (Placebo Comparator): Subjects will be treated with Placebo administered IM on Study Days 1, 29 and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PDA-002
  Arms: PDA-002 - 30X10^6 cells; PDA-002 -3x10^6 cells
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study PDA-002-DFU-003 is a Phase 2, multicenter, randomized, double blind, placebo-controlled, dose range finding study in subjects who have diabetic foot ulcer (DFU) with peripheral arterial disease (PAD). The study will enroll approximately 24 subjects. This study will investigate the hemodynamic effects, clinical efficacy, and safety of 3 monthly intramuscular (IM) injections of PDA-002 in subjects who have DFU with PAD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, at least 18 years of age or older at the time of signing the informed consent document.
2. Diabetes mellitus Type 1 or Type 2.
3. Diabetic foot ulcer with severity of Grade 1 (full thickness only) or Grade 2 on the Wagner Grading Scale of greater than one month duration which has not adequately responded to conventional ulcer therapy.
4. Subjects who meet one or more of the following criteria of arterial insufficiency in the foot with the index ulcer:

   1. Peripheral arterial disease with ABI ≥ 0.40 and ≤ 0.80 or TBI ≥0.30 and ≤ 0.65.
   2. Transcutaneous oxygen measurement between 20 to 40 mmHg.
5. No planned revascularization or amputation over the next 3 months after screening visit, in the opinion of the investigator.
6. Dosing should not begin until at least 14 days after a failed reperfusion intervention and at least 30 days after a successful reperfusion intervention

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study, at the discretion of the investigator.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he or she were to participate in the study, at the discretion of the investigator.
3. Pregnant or lactating females.
4. Subjects with a body mass index > 40 mg/m2 at Screening.
5. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 at Screening calculated using the Modification of Diet in Renal Disease Study equation or history of eGFR decline > 15 mL/min/1.73 m2 in the past year.
6. Untreated chronic infection or treatment of any infection with systemic antibiotics,including the ulcer site. Subject must be antibiotic free within 1 week prior to dosing with Investigational Product (IP).
7. Known osteomyelitis or infection or cellulitis at or adjacent to the index ulcer.
8. Limb pain at rest due to limb ischemia.
9. Uncontrolled hypertension (defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 180 mmHg during Screening at 2 independent measurements taken while subject is sitting and resting for at least 5 minutes).
10. Poorly controlled diabetes mellitus (hemoglobin A1c >12% or a screening serum glucose of ≥ 300 mg/dL).
11. Untreated proliferative retinopathy.
12. History of malignant ventricular arrhythmia, Canadian Cardiovascular Society (CCS) Class III-IV angina pectoris, myocardial infarction/PCI (percutaneous coronary intervention)/CABG (coronary artery bypass graft) in the preceding 6 months prior to signing the Informed Consent (ICF),pending coronary revascularization in the following 3 months, transient ischemic attack/cerebrovascular accident in the preceding 6 months, prior to signing the ICF and/or New York Heart Association [NYHA] Stage III or IV congestive heart failure.
13. Abnormal ECG: new right bundle branch block (BBB) ≥ 120 msec in the preceding 3 months prior to signing the ICF.
14. Uncontrolled hypercoagulation syndrome.
15. Life expectancy less than 2 years due to concomitant illnesses.
16. In the opinion of the investigator, the subject is unsuitable for cellular therapy.
17. History of malignancy within 5 years prior to signing the ICF except basal cell or squamous cell carcinoma of the skin or remote history of cancer now considered cured or positive Pap smear with subsequent negative follow-up.
18. History of hypersensitivity to any of the components of the product formulation (including bovine or porcine products, dextran 40, and dimethyl sulfoxide [DMSO]).
19. Subject has received an investigational agent -an agent or device not approved by the US Food and Drug Administration (FDA) for marketed use in any indication- within 90 days (or 5 half-lives, whichever is longer) prior to treatment with study therapy or planned participation in another therapeutic study prior to the completion of this study.
20. Subject has received previous investigational gene or cell therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Ankle-brachial Index (ABI) | Approximately 1 year
  The ankle brachial index is the ratio of the measurement of the blood pressure in the ankle and the arm.
Transcutaneous oxygen measurement (TCOM) | Approximately 1 year
  Transcutaneous oxygen measurement measures the oxygen flow in vessels beneath the skin surface

SECONDARY OUTCOMES:
Adverse Events (AEs) | Approximatly 1 year
  Number of participants with adverse events
Ulcer closure | Approximatly 1 year
  Ulcer closure is defined as skin closure of the index ulcer without drainage or need for dressing.
Complete wound closure of the index ulcer | Approximatly 1 year
  Complete wound closure is defined as closure of the index ulcer and retaining wound closure for the subsequent 4 weeks.
Number of ulcers | Approximatly 1 year
  The total number of non index ulcers will be collected
Size of ulcers | Approximatly 1 year
  The area of each ulcer will be collected.
50% closure of the index ulcer | Approximatly 1 year
  The time to when the ulcer has closed 50 % will be collected.
Time to major amputation (above the ankle) of treated leg | Approximatly 1 year
  The time to a major amputation (above the ankle) will be collected.
Wagner Grading Scale | Approximatly 1 year
  The extent of the ulcer will be collected using a standard scale for ulcer assessment.
Rutherford Criteria | Approximately 1 year
  The extent of symptoms associated with decreased limb perfusion will be collected using a standard scale.
Leg Rest Pain Score Visual Analog Scale (VAS) | Approximately 1 year
  Pre and Post treatment Limb Pain level will be assessed using a VAS
Patient Global Impression of Change in Neuropathy (PGICN) | Approximately 1 year
  Subjects will be assessed for symptoms of diabetic neuropathy using a standard scale.

CONTACTS AND LOCATIONS:
Overall Officials: Monica E Luchi, MD, Study Director — Celularity Incorporated
Locations (1):
- University of Pennsylvania Health Systems, Philadelphia, Pennsylvania, United States